CLINICAL TRIAL: NCT04316936
Title: Evaluation of Efficacy in the Resolution of Post-Operative Inflammation and Pain in Patients Receiving Omidria and Dexycu, or Omidria and Dextenza Compared to Topical Prednisolone Acetate 1% Following Cataract Surgery
Brief Title: Omidria and Dexycu, or Omidria and Dextenza Compared to Topical Prednisolone Acetate 1% Following Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Silverstein Eye Centers (Other)
Collaborators: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2020-03-17; First posted 2020-03-20 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Cataract Surgery
Keywords: Dextenza; intracanalicular dexamethasone; dexamethasone ophthalmic insert; Dexycu; Omidria
MeSH Terms: interventions — Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to 1 of 3 groups (1:1:1), each with a sample size of 25 (total n=75). Group 1 will receive DEXYCU + Omidria (Omidria = ketorolac + phenylephrine), group 2 will receive DEXTENZA + Omidria, and group 3 will receive prednisolone acetate + Omidria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Omidria + Dextenza (dexamethasone ophthalmic insert) 0.4mg (Experimental): Omidria (= ketorolac + phenylephrine) and intracanalicular dexamethasone insert (punctal plug)
  Interventions: Drug: Omidria; Drug: Dextenza (dexamethasone ophthalmic insert) 0.4mg
- Omidria + Dexycu (Experimental): Omidria (= ketorolac + phenylephrine) and intraocular dexamethasone suspension
  Interventions: Drug: Omidria; Drug: Dexycu, 9% Intraocular Suspension
- Omidria + Prednisolone Acetate 1% (Active Comparator): Omidria (= ketorolac + phenylephrine) and topical prednisolone acetate ophthalmic drops
  Interventions: Drug: Omidria; Drug: Prednisolone Acetate 1%

INTERVENTIONS:
Drug: Omidria — phenylephrine 1% and ketorolac 0.3% intraocular solution
Drug: Dextenza (dexamethasone ophthalmic insert) 0.4mg — intracanalicular dexamethasone insert
  Arms: Omidria + Dextenza (dexamethasone ophthalmic insert) 0.4mg
Drug: Dexycu, 9% Intraocular Suspension — dexamethasone intraocular suspension
  Arms: Omidria + Dexycu
Drug: Prednisolone Acetate 1% — standard postoperative ophthalmic drop regimen
  Arms: Omidria + Prednisolone Acetate 1%

SUMMARY:
This research will evaluate the efficacy of Omidria and Dexycu, Omidria and Dextenza, and Omidria and prednisolone acetate 1% in the resolution of post-operative inflammation and pain following cataract surgery.

DETAILED DESCRIPTION:
Prospective, randomized trial where patients will be randomly assigned to 1 of 3 groups, each with a sample size of 25 (total n=75). Group 1 will receive DEXYCU + Omidria (Omidria = ketorolac + phenylephrine), group 2 will receive DEXTENZA + Omidria, and group 3 will receive prednisolone acetate + Omidria. Each of the drug combinations used in each of the 3 groups is standard of care, FDA approved, and will be used on label. 1:1:1, n=75 with 25 subjects assigned to each of the 3 groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older, undergoing routine, uncomplicated cataract surgery.

Exclusion Criteria:

* Any history of corneal dystrophy, corneal surgery within 6 months of cataract surgery, previous intraocular surgery, any concomitant eye drop use besides artificial tears, previous ocular trauma, or a history of treated glaucoma. No additional procedures can be done at the time of cataract surgery (e.g., stent placement, endo-laser, etc.), but femto-second laser-assisted surgery is permitted.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Resolution of anterior chamber inflammation | Assessed at day 8 post-operatively
  The primary efficacy end point is the complete resolution of anterior chamber inflammation (cell and flare). This is a non-contact, non-invasive test performed by the physician using a slit lamp. The evaluation requires less than one minute.
Resolution of anterior chamber inflammation | Assessed at day 15 post-operatively
  The primary efficacy end point is the complete resolution of anterior chamber inflammation (cell and flare). This is a non-contact, non-invasive test performed by the physician using a slit lamp. The evaluation requires less than one minute.
Resolution of anterior chamber inflammation | Assessed at day 30 post-operatively
  The primary efficacy end point is the complete resolution of anterior chamber inflammation (cell and flare). This is a non-contact, non-invasive test performed by the physician using a slit lamp. The evaluation requires less than one minute.

SECONDARY OUTCOMES:
Resolution of postoperative pain | Assessed at day 1 post-operatively
  The secondary efficacy endpoint is the elimination of post-operative pain per a subjective, standardized scale. Post-operative pain as measured on a scale from 0-10 (ocular pain assessment).
Resolution of postoperative pain | Assessed at day 8 post-operatively
  The secondary efficacy endpoint is the elimination of post-operative pain per a subjective, standardized scale. Post-operative pain as measured on a scale from 0-10 (ocular pain assessment).

OTHER OUTCOMES:
Optical Coherence Tomography (OCT) | Assessed pre-operatively and 1 month post-operatively
  OCT is a non-contact, non-invasive test that takes less than a minute to perform. All that is required of the patient is that they sit still and look at a fixation light while the machine takes a picture. No eye drops or any other intervention are required. OCT scanning will provide an image of the deep layers of the retina and will be used to determine macular thickness measurement (macular thickness has been correlated to changes in contrast sensitivity) before and 30 days following surgery. .
Contrast sensitivity testing | Assessed pre-operatively, and at 15 days and 30 days post-operatively
  This test is non-contact, non-invasive and used to distinguish between finer and finer increments of light versus dark. The patient simply looks at a chart similar to the Snellen Eye Chart and distinguishes lighter shades from darker shades. The test is performed in less than one minute.
Best corrected visual acuity | Assessed pre-operatively, and at 15 days and 30 days post-operatively
  ETDRS chart at 4m
Optical Coherence Tomography (OCT) | Assessed pre-operatively and 1 month post-operatively
  OCT is a non-contact, non-invasive test that takes less than a minute to perform. All that is required of the patient is that they sit still and look at a fixation light while the machine takes a picture. No eye drops or any other intervention are required. OCT scanning will provide an image of the deep layers of the retina and will be used to evaluate for the presence of cystoid macular edema before and 30 days following surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Silverstein Eye Centers, Kansas City, Missouri, United States